CLINICAL TRIAL: NCT05520255
Title: 18F-PSMA-1007 PET/CT in Prostate Cancer - Access Trial 2022 to 2028
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CC-22-0204
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Two-centre prospective cohort phase III study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-PSMA-1007 (Experimental): 18F-PSMA-1007, 4 MBq/kg (max 400 MBq; +/- 15%), intravenous, single dose
  Interventions: Drug: 18F-PSMA-1007

INTERVENTIONS:
Drug: 18F-PSMA-1007 — 18F-PSMA-1007 intravenous injection

SUMMARY:
A two-centre prospective cohort phase III study of 18F-PSMA-1007 PET/CT imaging in specific patient populations:

1. Adults patients (≥18 years old) with a history of radical prostatectomy for treatment of prostate cancer, and a serum prostate specific antigen (PSA) ≥ 0.2 mcg/L
2. Adult patients with a history of radiotherapy, cryotherapy, or brachytherapy for treatment of prostate cancer, and a serum PSA progressively rising to ≥ 2 mcg/L (minimum two samples) OR a serum PSA doubling time of < 9 months
3. Adult patients with a history of biopsy-proven prostate cancer and high-risk features for metastatic disease prior to treatment with radical prostatectomy, radiotherapy, cryotherapy, or brachytherapy. High-risk features include a Gleason score ≥ 7, serum PSA ≥ 20 mcg/L, OR minimum clinical T-stage T2c
4. Adult patients who do not meet criteria 1-3 but in whom a 18F-PDAM-1007 PET/CT scan is expected to provide clinical benefit as determined by a Urologist, Radiation Oncologist, Medical Oncologist, or Nuclear Medicine physician (licensed in Alberta)

The safety of the investigational 18F-PSMA-1007 tracer will be evaluated in 3 ways:

1. The participant will be screened for adverse effects immediately post-injection
2. The participant will be screened for adverse effects immediately after the scan (approximately 2.5 hours after tracer injection)
3. The participant will be provided an information sheet and contact information for self-reporting of any delayed adverse events (1-7 days post injection)

The incidence of and activity of non-specific bone lesions will be quantified and evaluated as follows:

1. All lesions categorized as non-specific bone lesions (PSMA-1007 SUVmax > 2.5 but no corresponding lesion on CT) will be recorded
2. The SUVmax and anatomic location will be recorded for each lesion (max 5 per participant)
3. Recorded lesions will be evaluated a minimum of 1 year post-scan to determine whether they are benign or malignant based on previously published reference standard criteria (Arnfield et al., 2021)
4. Equivocal lesions will be considered unevaluable and will be excluded from assessment of accuracy

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants (≥ 18 years old) with a history of radical prostatectomy for treatment of prostate cancer, and a serum prostate specific antigen (PSA) ≥ 0.2 mcg/L
2. Adult participants with a history of radiotherapy, cryotherapy, or brachytherapy for treatment of prostate cancer, and a serum PSA progressively rising to ≥ 2 mcg/L (minimum two samples) OR a serum PSA doubling time of < 9 months
3. Adult participants with a history of biopsy-proven prostate cancer and high-risk features for metastatic disease prior to treatment with radical prostatectomy, radiotherapy, cryotherapy, brachytherapy, or other similar therapy. High-risk features include a Gleason score ≥ 7, serum PSA ≥ 20 mcg/L, OR minimum clinical T-stage T2c
4. Adult patients who do not meet criteria 1-3 but in whom a 18F-PSMA-1007 PET/CT scan is expected to provide clinical benefit as determined by a Urologist, Radiation Oncologist, Medical Oncologist, or Nuclear Medicine physician (licensed in Alberta)

Exclusion Criteria:

1. Unable to obtain consent
2. Weight > 225 kg (weight limit of PET/CT scanners)
3. Unable to lie flat for 30 minutes to complete the PET/CT imaging session
4. Lack of intravenous access
5. History of allergic reaction to 18F-PSMA-1007
6. Residence outside the Province of Alberta, Northwest Territory, or Yukon Territory (Canada)
7. Less than 18 years old

NOTE: Androgen deprivation therapy (ADT) is NOT a contraindication to participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Safety - immediate | Immediately after tracer injection
  The participant will be screened for adverse effects immediately post-injection
Safety - post scan | 2.5 hours after tracer injection
  The participant will be screened for adverse effects immediately after the scan (approx 2.5 hours after injection).
Safety - delayed | 1-7 days after tracer injection
  The participant will be provided information to contact the study team to self-report and delayed adverse events (1-7 days post-injection)
Non-specific bone lesion assessment (NSBLs) | 1 year after tracer injection
  SUVmax and anatomic location of NSBLs (max 5 per participant) will be compared to a reference standard 1 year after tracer injection

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No